CLINICAL TRIAL: NCT02408406
Title: PatientCareAnywhere: Patient Support and Empowerment Across the Care Continuum
Brief Title: PatientCareAnywhere Internet-Based Software in Improving Communication and Education in Patients With Cancer and Their Healthcare Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15025; NCI-2015-00554 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 115352; 15025 (Other: City of Hope Comprehensive Cancer Center); R44CA192588 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Bladder Carcinoma; Breast Carcinoma; Colorectal Carcinoma; Lung Carcinoma; Malignant Female Reproductive System Neoplasm; Malignant Neoplasm
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (PatientCareAnywhere program system) (Experimental): Patients are encouraged to use the PatientCareAnywhere program at least once weekly either in the clinic or at home. Patients receive reminder emails after 1 week of inactivity. If patients indicate they are experiencing moderate to severe symptoms, an alert message is sent to at least 1 member of the patient's support team along with a list of expected response times.
  Interventions: Other: Communication Intervention; Other: Educational Intervention; Other: Internet-Based Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients receive usual care, including a one-time use of SupportScreen, a touchscreen questionnaire system that identifies patient issues before appointments, at the clinic during the first treatment consultation after diagnosis. Consultation, printed education materials, and specialist referrals may be generated based on SupportScreen responses.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Use PatientCareAnywhere system
  Arms: Arm I (PatientCareAnywhere program system)
Other: Educational Intervention — Use PatientCareAnywhere system
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (PatientCareAnywhere program system)
Other: Internet-Based Intervention — Use PatientCareAnywhere system
  Arms: Arm I (PatientCareAnywhere program system)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This partially randomized pilot clinical trial develops and studies a software program, called PatientCareAnywhere, to see whether it can help patients communicate with their doctors and other healthcare providers, and educate themselves about their cancer and treatment options. A program that can help patients learn about their cancer and treatment options, and allows the patient's healthcare providers to receive their questionnaire results, may help patients identify and get help to treat their symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Solicit stakeholder feedback on expected system functions, perceived usefulness and impacts, and potential adoption barriers via 10 focus groups. (Human Subjects [HS], Phase I) II. Develop the software prototype using an iterative user-centered design process and leverage the technical design and components from an existing clinic-based biopsychosocial screening tool and an existing patient portal solution as well as the patient education contents from City of Hope (COH). (Phase I) III. Conduct two usability tests with 24 subjects each to evaluate the usability, usefulness, and acceptability of the prototype system developed in Aim 2. (HS, Phase I) IV. Conduct a 50-subject pilot evaluation study to demonstrate the feasibility of our technical solution and our Phase II randomized controlled trial protocol design. (HS, Phase I) V. Enhance the software system to add more administrative/customization features and to expand the education contents to cover more cancer types and treatment options. (Phase II) VI. Conduct a 2-year 516-subject randomized control trial to test the effectiveness hypothesis. (HS, Phase II)

OUTLINE:

FOCUS GROUPS: Ten, 90-minute focus group sessions are conducted, composed of patients; caregivers, friends, and family members; cancer treatment professionals; supportive care professionals and community support professionals. Sessions address what functions participants expect to see in the program, what benefits are expected, and any expected barriers for using the program.

USABILITY EVALUATION (DESIGN-ORIENTED & METRIC-ORIENTED): Patients, caregivers, and clinical care/support professionals in each type of evaluation undergo a 60-minute one-on-one session in which they are assigned tasks to complete using the system, and an observer records how the tasks are completed. Participants are also requested to talk aloud while performing the task. Participants in the metric-oriented evaluation respond to usability and usefulness questionnaires.

PILOT STUDY & RANDOMIZED CONTROLLED TRIAL: Patients are randomized to 1 of 2 arms.

ARM I (INTERVENTION GROUP): Patients are encouraged to use the PatientCareAnywhere program at least once weekly either in the clinic or at home. Patients receive reminder emails after 1 week of inactivity. If patients indicate they are experiencing moderate to severe symptoms, an alert message is sent to at least 1 member of the patient's support team along with a list of expected response times.

ARM II (CONTROL GROUP): Patients receive usual care, including a one-time use of SupportScreen, a touchscreen questionnaire system that identifies patient issues before appointments, at the clinic during the first treatment consultation after diagnosis. Consultation, printed education materials, and specialist referrals may be generated based on SupportScreen responses.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I AIM 1 (STAKEHOLDER INPUT)
* PHASE I AIM 1: Malignant diagnosis in any cancer type at any stage
* PHASE I AIM 1: Receiving any type of cancer treatment
* PHASE I AIM 1: Life expectancy of at least six months
* PHASE I AIM 1: Current outpatient status
* PHASE I AIM 1: Fluent in English
* PHASE I AIM 1: Internet access at home
* PHASE I AIM 3.1 (EVALUATION STUDY)
* PHASE I AIM 3.1: Malignant diagnosis in any cancer type at any stage
* PHASE I AIM 3.1: Receiving any type of cancer treatment
* PHASE I AIM 3.1: Life expectancy of at least six months
* PHASE I AIM 3.1: Current outpatient status
* PHASE I AIM 3.1: Fluent in English
* PHASE I AIM 3.1: Internet access at home
* PHASE I AIM 3.2 (PILOT STUDY)
* PHASE I AIM 3.2: Malignant diagnosis in breast, gynecologic (GYN), genitourinary (GU) cancer at any stage
* PHASE I AIM 3.2: Receiving surgery and/or chemotherapy treatment
* PHASE I AIM 3.2: Life expectancy of at least six months
* PHASE I AIM 3.2: Current outpatient status (participation will be suspended during hospitalization)
* PHASE I AIM 3.2: Fluent in English
* PHASE I AIM 3.2: Internet access at home
* PHASE II AIM 2 (RANDOMIZED CONTROLLED TRIAL)
* PHASE II AIM 2: Malignant diagnosis of breast, lung, or colorectal cancer at any stage
* PHASE II AIM 2: Receiving any type of cancer treatment
* PHASE II AIM 2: Life expectancy of at least six months
* PHASE II AIM 2: Current medical oncology outpatient status (participation will be suspended during hospitalization)
* PHASE II AIM 2: Fluent in English
* PHASE II AIM 2: Internet access at home

Exclusion Criteria:

* PHASE I AIM 1 (STAKEHOLDER INPUT) EXCLUSION
* PHASE I AIM 1: Clinical evidence of cognitive or psychological impairment
* PHASE I AIM 1: Prisoners and pregnant women
* PHASE I AIM 3.1 (EVALUATION STUDY) EXCLUSION
* PHASE I AIM 3.1: Clinical evidence of cognitive or psychological impairment
* PHASE I AIM 3.1: Prisoners and pregnant women
* PHASE I AIM 3.2 (PILOT STUDY) EXCLUSION
* PHASE I AIM 3.2: Clinical evidence of cognitive or psychological impairment
* PHASE I AIM 3.2: Prisoners and pregnant women
* PHASE I AIM 3.2: Currently participating in other psychosocial studies
* PHASE II AIM 2 (RANDOMIZED CONTROLLED TRIAL) EXCLUSION
* PHASE II AIM 2: Clinical evidence of cognitive or psychological impairment
* PHASE II AIM 2: Prisoners and pregnant women
* PHASE II AIM 2: Currently participating in other psychosocial studies

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-07-07 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-General (FACT-G) scores | Up to 6 months
  Separate analysis will be carried out for the per-protocol (PP) population and intent-to-treat (ITT) population. For the PP population, a repeated measures analysis of variance will be employed. In this model, FACT-G scores are the response variables. Time, patient group and their interaction are the predictors. For the ITT population, a random effect model will be fitted to the data. The model can also adjust for covariates of potential interests. Exploratory assessments may also include effects of other variables of interest, such as demographic and baseline values.

SECONDARY OUTCOMES:
Change in self-efficacy as measured by the revised Chronic Disease Self-Efficacy Scale | Baseline to up to 6 months
  Analysis steps follow those for the primary outcome.
Change in health resource utilization | Baseline to up to 6 months
  Measured by number of unplanned hospitalizations, emergency room visits, intensive care unit stays, diagnostic tests, and clinic no-shows. Analysis steps follow those for the primary outcome.

OTHER OUTCOMES:
Individual patient changes in Functional Assessment of Cancer Therapy-General (FACT-G) total scores | Baseline to 3 months
  Categorized as improved (+ 10% or higher compared to baseline), unchanged (-9.9% to +9.9%), or declined (- 10% or lower compared to baseline). Missing data will be accounted for using the last-observation-carried-forward value. The proportion of patients in each category will be calculated per patient group. Differences in category proportions per patient group will be investigated via ordinal logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Clark, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Baik SH, Clark K, Sanchez M, Loscalzo M, Celis A, Razavi M, Yang D, Dale W, Haas N. Usability and Preliminary Efficacy of an Adaptive Supportive Care System for Patients With Cancer: Pilot Randomized Controlled Trial. JMIR Cancer. 2024 Jul 10;10:e49703. doi: 10.2196/49703. PMID 38986134